CLINICAL TRIAL: NCT05319964
Title: Comparison of Anti-gravity Treadmill Training and Traditional Treadmill Training in Patients With Moderate to Severe Knee Osteoarthritis
Brief Title: Anti-gravity Treadmill Training in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuğba Atan, MD, Assoc. Prof, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-21-1004
Record Dates: First submitted 2022-03-28; First posted 2022-04-11 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anti-gravity treadmill (Experimental): Patients in all three study groups will receive hot pack, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound 3 days a week for 8 weeks.
  Participants were provided 30 minutes anti-gravity treadmill sessions including a 5 minutes warm - up and cool - down period for each session, 3 days a week, for 8 weeks
  Interventions: Behavioral: Anti-gravity treadmill
- conventional treadmill (Active Comparator): Patients in all three study groups will receive hot pack, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound, 3 days a week for 8 weeks.
  The moderate-intensity aerobic exercise program will be performed for 30 minutes at an intensity of 65-80% of the maximum heart rate, consisting of a 5-minute warm-up and cool-down period.
  Interventions: Behavioral: Conventional treadmill
- Control (Other): Patients in all three study groups will receive hot pack, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound 3 days a week for 8 weeks
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Anti-gravity treadmill — Patients in all three study groups will receive hot pack, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound, 3 days a week for 8 weeks.
  Participants were provided 30 minutes anti-gravity treadmill sessions including a 5 minutes warm - up and cool - down period for each session, 3 days a week, for 8 weeks
  Arms: anti-gravity treadmill
Behavioral: Conventional treadmill — Patients in all three study groups will receive hot pack, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound 3 days a week for 8 weeks.
  The moderate-intensity aerobic exercise program will be performed for 30 minutes at an intensity of 65-80% of the maximum heart rate, consisting of a 5-minute warm-up and cool-down period.
  Arms: conventional treadmill
Behavioral: Control — Patients in all three study groups will receive hot pack, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound 3 days a week for 8 weeks.
  Arms: Control

SUMMARY:
The aim of this study is to compare anti-gravity treadmill training with traditional treadmill training in patients with moderate to severe knee osteoarthritis.

DETAILED DESCRIPTION:
Patients with moderate to severe OA have persistent pain that significantly affects their functional status, activity participation, and quality of life. As with mild OA, non-pharmacological interventions that focus on education, exercise, and weight management are first-line treatments for patients with moderate to severe knee OA.

Exercise is recommended for all patients with moderate to severe knee OA to reduce pain and protect the joint. A meta-analysis showed that exercise has beneficial effects on pain, even in patients with severe disease and awaiting total knee replacement.Therefore, the objective of this study was to compare the effects of anti-gravity treadmill training and traditional treadmill training on pain levels, quality of life and functional capacity in patients with moderate and severe knee osteoarthritis.

In addition, it was aimed to compare the compliance of the patients to aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 50 and ≤ 75 years old
* Patients with a diagnosis of knee OA in at least one knee according to the classification criteria of the American College of Rheumatology
* Patients with Kellgren-Lawrence (K-L) knee OA staging III to IV
* Patients reporting knee pain on most days of the past month
* Patients with stable medical and psychological status
* Patients willing to participate in the study

Exclusion Criteria:

Patients with serious cardiovascular, pulmonary, neurological disease or other musculoskeletal problems (inflammatory rheumatic disease, active synovitis, severe low back pain, hip/knee joint replacement or other hip/knee-related trauma, fracture, or surgery) that impair walking

* Patients with a history of corticosteroid injection to the knee in the last 3 months
* Patients who have received opioid analgesics or systemic corticosteroids in the last 3 months
* Patients who have undergone any exercise program or physical therapy program for the lower extremities in the last 3 months
* Patients with severe vision, hearing and language problems
* Patients with a body mass index ≥35 kg /m²

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain (VAS-pain) | Baseline - Change from Baseline at 4 weeks - Change from Baseline at 8 weeks
  Pain intensity will be evaluated with a visual analog scale (0-10mm) that has proven validity and reliability to measure musculoskeletal pain.

SECONDARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) Score | Baseline - Change from Baseline at 4 weeks - Change from Baseline at 8 weeks
  It measures knee pain, stiffness, and physical function. Scores for each subscale are summed with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. The sum of the scores of the three subscales gives the WOMAC score. High scores are associated with more pain, stiffness, and dysfunction, while low scores indicate well-being.
Six-minute walk test (6MWT) | Baseline - Change from Baseline at 4 weeks - Change from Baseline at 8 weeks
  The 6 Minute Walk Test is a submaximal exercise test that usually corresponds to 80% of a person's maximum heart rate and is used to evaluate functional capacity and treatment response.
Femoral cartilage thickness measurement with ultrasound | Baseline - Change from Baseline at 4 weeks - Change from Baseline at 8 weeks
  Distal femoral cartilage thickness will be evaluated by the same investigator, blinded to the patient treatment groups, using an ultrasound device with a 7.5-12 MHz linear transducer (LOGIQ 7 Pro; GE Yokogawa Medical System, Tokyo, Japan) available in our clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Therapy and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atan T, Bildik YE, Demir Y, Guzelkucuk U, Tan AK. Comparison of anti-gravity treadmill training and traditional treadmill training in patients with moderate to severe knee osteoarthritis: A randomized controlled trial. Ir J Med Sci. 2025 Feb;194(1):125-136. doi: 10.1007/s11845-024-03836-w. Epub 2024 Nov 1. PMID 39482393